CLINICAL TRIAL: NCT01235624
Title: Autosomal Dominant Retinitis Pigmentosa: Prevalence of Known Genes Identification of New Loci / Genes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UF 8300; 2008-A01238-47
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Autosomal Dominant Retinitis Pigmentosa
Keywords: Autosomal dominant retinitis pigmentosa; Rare disease; Genetics
MeSH Terms: conditions — Rare Diseases | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patient (Other): Patient suffering of adRP that accept to participate at this study have a blood prelevement for genetic analysis (intervention)
  Interventions: Genetic: genetic analysis

INTERVENTIONS:
Genetic: genetic analysis

SUMMARY:
Identify new genes responsible for autosomal dominant retinitis pigmentosa (ADRP), one of the most common causes of hereditary diseases of the retina, and thus better understand the mechanisms involved of the disease."

DETAILED DESCRIPTION:
Two hundred and fifty samples from unrelated patients, from which 150 were provided by the national reference center of rare disease in Montpellier and 100 recruited in the 9 participating centers over a period of two years."To identify the missing genes, we proceed in two steps. A first step in selecting families negative for the 8 major genes genes, by systematic sequencing of exons most frequently involved. A second step in finding new loci / genes by locus exclusion using microsatellite markers and SNP genotyping.

ELIGIBILITY:
Inclusion Criteria:

* retinitis pigmentosa diagnosed
* Autosomal dominant transmission diagnosed
* Aged from 5 to 80 years
* Informed consent
* Affiliated or benefit from an insurance regimen

Exclusion Criteria:

-

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1161 (Actual)
Dates: Start 2009-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
identification of unknown loci and genes responsible of Autosomal dominant retinitis pigmentosa (adRP) | for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: christian HAMEL, Pr Ph.D, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; José-Alain SAHEL, Pr, Study Chair — § Centre hospitalier national d'ophtalmologie des XV-XX, Paris,FRANCE; Jean Louis DUFIER, Pr, Study Chair — Hopital Necker enfants-malades,Paris,FRANCE; Hélène DOLLFUS, Pr, Study Chair — CHU de STRASBOURG, FRANCE; sylvie ODENT, Pr, Study Chair — CHU de RENNES Unité INSERM 598,Paris,FRANCE; Sabine DEFOORT- DHELEMMES, Ph.D, Study Chair — CHRU de LILLE,FRANCE; Michel WEBER, Pr, Study Chair — CHU de NANTES,FRANCE; Xavier ZANLONGH, Ph.D, Study Chair — CLINIQUE SOURDILLE, NANTES,France; Laurence LO OLIVIER-FAIVRE, PH, Principal Investigator — Centre génétique Médicale - Children Hospital of DIJON
Locations (1):
- CHRU Montpellier, Montpellier, France

REFERENCES:
- [Result] Audo I, Manes G, Mohand-Said S, Friedrich A, Lancelot ME, Antonio A, Moskova-Doumanova V, Poch O, Zanlonghi X, Hamel CP, Sahel JA, Bhattacharya SS, Zeitz C. Spectrum of rhodopsin mutations in French autosomal dominant rod-cone dystrophy patients. Invest Ophthalmol Vis Sci. 2010 Jul;51(7):3687-700. doi: 10.1167/iovs.09-4766. Epub 2010 Feb 17. PMID 20164459